CLINICAL TRIAL: NCT03767465
Title: Treatment With Immunological Checkpoint Inhibitors of HIV-infected Subjects With Cancer
Acronym: PembroHIV
Status: Completed | Type: Observational
Sponsor: IrsiCaixa (Other)
Responsible Party: Sponsor
Other Study IDs: PembroHIV
Record Dates: First submitted 2018-12-03; First posted 2018-12-06 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: HIV Infection; Cancer
Keywords: HIV; Cancer; Checkpoint inhibitors; HIV reservoir; Immunity
MeSH Terms: conditions — HIV Infections; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Criopreserved peripheral blood mononuclear cells (PBMCs) Frozen plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- PembroHIV: HIV-infected subjects with advanced melanoma or other oncological conditions in which the use of immunological checkpoint inhibitors is clinically indicated

SUMMARY:
It has been reported that peripheral and lymph node resident Cluster of Differentiation 4 (CD4)+ T cells expressing Programmed cell death protein 1 (PD-1) contribute to Human Immunodeficiency Virus (HIV) persistence during Antiretroviral Therapy (ART). In HIV-infected individuals, PD-1 expression on CD4+ T cells correlates with HIV disease progression, and loss of HIV-specific CD4+ T cell function can be reversed in vitro by PD-1 blockade. There are only a limited number of case reports describing the evolution of HIV-infected patients with concurrent oncological disease treated with immunological checkpoint inhibitors. However, this case provides very limited information on the effect of pembrolizumab on the HIV reservoir. Here, the investigators aim at describing changes in the HIV reservoir and in the HIV-specific immunity in HIV-infected patients on ART who receive immunological checkpoint inhibitors for the treatment of cancer, especially for metastatic melanoma.

DETAILED DESCRIPTION:
Long-lived latently infected resting CD4+ T cells are the main reason why current antiretroviral therapy (ART) is unable to cure HIV infection. Recent work has suggested that the expression of immune checkpoint markers, such as the programmed death-1 (PD1) or the cytotoxic T-lymphocyte antigen 4 (CTL-4), may play a role in viral persistence on ART via either suppression of virus transcription and/or reduced HIV-specific T cell activity, but the in vivo role of immune checkpoint markers in HIV persistence on ART is not clear.

Immunological checkpoint inhibitors are humanized monoclonal Immunoglobulin G (IgG) antibodies directed against several cell surface receptors, including PD-1 that inhibits binding of PD-1, expressed on activated T cells to its ligands PD-L1, overexpressed on certain cancer cells, and PD-L2, which is primarily expressed on antigen presenting cells. Activated PD-1 negatively regulates T-cell activation and plays a key role in tumor evasion from host immunity antigen presenting cells. Immunological checkpoint inhibitors can also target CTL-4, which is constitutively expressed in Treg cells but only upregulated in conventional T cells after activation, a phenomenon which is particularly notable in cancers. These drugs are used to treat oncology diseases, including metastatic melanoma, and have been associated with multiple changes in immune function thought to enhance antitumor T cell function.

This exploratory study will include HIV-infected subjects with advanced melanoma or other oncological conditions in which the use of immunological checkpoint inhibitors is clinically indicated. The study is conceptually observational as the patients will be in regular clinical treatment with immunological checkpoint inhibitors for oncological conditions.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected subjects with advanced melanoma or other oncological conditions in which the use of immunological checkpoint inhibitors is clinically indicated

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: HIV-infected subjects with advanced melanoma or other oncological conditions in which the use of immunological checkpoint inhibitors is clinically indicated
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Quantification of total HIV DNA | At the end of recruitment (up to one year after inclusion)
  Measurement of HIV viral latency by quantification of total HIV DNA in purified CD4+ T cells, using digital droplet PCR (ddPCR)
Quantification of cell-associated HIV RNA | At the end of recruitment (up to one year after inclusion)
  Measurement of viral transcription by quantification of cell-associated unspliced HIV RNA in purified CD4+ T cells, using ddPCR
Quantification of ultrasensitive HIV viral load | At the end of recruitment (up to one year after inclusion)
  Measurement of ultrasensitive viremia in plasma using single copy assay
Analysis of changes in HIV-specific cellular responses | At the end of recruitment (up to one year after inclusion)
  Changes in the ability of Peripheral Blood Mononuclear Cells (PBMCs) to release Interferon gamma (IFNγ) in response to viral antigen stimulation (ELISPOT assay).
Analysis of changes in immune-phenotype of cellular populations | At the end of recruitment (up to one year after inclusion)
  Study of changes in multiple cell membrane markers related with cell function, including T-cell activation and proliferation, T-cell exhaustion, T-cell subpopulations and release of specific cytokines in response to HIV stimuli (multicolor flow cytometry).
Analysis of changes in HIV inhibition capacity in vitro | At the end of recruitment (up to one year after inclusion)
  Changes in the ex vivo ability of cluster of differentiation 8 (CD8)+ T cells to inhibit superinfected autologous CD4+ T cells (virus inhibition assay).
Supervision of changes on the standard blood analysis for oncologic follow-up | At the end of recruitment (up to one year after inclusion)
  Blood analysis will be revised for oncologic follow-up
Analysis of changes in imaging of the oncological focus | At the end of recruitment (up to one year after inclusion)
  Positron Emission Tomography (PET) scan will be analyzed for oncologic follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Javier Martinez-Picado, PhD, Principal Investigator — IrsiCaixa
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided